CLINICAL TRIAL: NCT06491316
Title: Long Term Results of Cross-leg Free Vascularized Fibular Transfer for Reconstruction of Complex Post-traumatic Tibial Bone Defects: a Case Series Study
Brief Title: Results of Cross-leg Free Vascularized Fibular Graft
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammad Saad, Demonstrator at Orthopedics and Trauma surgery department, Assiut university hospital, Assiut University
Other Study IDs: Results of Cross-leg FVFG
Record Dates: First submitted 2023-03-20; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Tibial Fractures
Keywords: Cross-leg flap; Vascularized fibular transfer; Open grade III tibial fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the new technique of cross-leg vascularized fibular graft for reconstruction of post-traumatic long tibial bone defects in terms of restoring normal anatomy and function of the traumatized limb in a series of cases admitted in Assiut University hospital, Orthopedics and trauma surgery department.

DETAILED DESCRIPTION:
Reconstruction of post-traumatic long tibial bone defects is still a major therapeutic challenge faced by orthopaedic surgeons on both anatomical and functional concerns, and it is usually associated with significant long-term morbidity. Historically, Amputation was the treatment of choice for long tibial bone defects because of difficulty of reconstructove management of such cases. Over the last few decades, Limb salvage procedures have been developed. During the second world war, massive cancellous bone autograft has been the preferred treatment. But traditional bone graft procedures in many cases may be limited by uncontrollable graft resorption. To overcome this disadvantage different management options have been developed to address bone defects of various lengths as vascularized fibular grafts, Ilizarov technique using bifocal or trifocal bone transport, acute limb shortening and masquelet procedure. However, In some cases long bone defects are associated with extensive soft tissue lacerations together with poor ipsilateral blood supply. For those cases previous surgical options are associated with many complications and may end up with failure of reconstruction and amputation, in this situation cross-leg vascularized fibular graft may be a good treatment option because it can provide a blood supply away from that of the extensively traumatized limb.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were admitted into Assiut University Hospital, Orthopedics and Trauma Surgery department with big tibial bone defects ranging from 12 cm to 26 cm, associated with extensive soft tissue damage and poor ipsilateral blood supply confirmed by CT angiography and treated with cross-leg free vascularized fibular graft.

Exclusion Criteria:

* Patients with bilateral extensive soft tissue damage and poor blood supply.
* Patients with medical conditions preventing them from general anesthesia for long periods (>10 hours).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases who were presented to Assiut University Hospital, Orthopedics and Trauma Surgery department with big tibial bone defects ranging from 12 cm to 26 cm, associated with extensive soft tissue damage and poor ipsilateral blood supply confirmed by CT angiography and treated with cross-leg free vascularized fibular graft and are presented recently for achieving long term results assessment.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of cases of Flap survival | 6 weeks from operation
  Flap intake and vascularization without necrosis
Number of cases of Bone healing | 1 year from operation
  Radiological evaluation

SECONDARY OUTCOMES:
Number of cases with accepted Limb alignment | 1 year
  Long film x-ray of both lower limbs to assess bone alignment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Watson JT, Anders M, Moed BR. Management strategies for bone loss in tibial shaft fractures. Clin Orthop Relat Res. 1995 Jun;(315):138-52. PMID 7634662
- [Background] Weinberg H, Roth VG, Robin GC, Floman Y. Early fibular bypass procedures (tibiofibular synostosis) for massive bone loss in war injuries. J Trauma. 1979 Mar;19(3):177-81. doi: 10.1097/00005373-197903000-00008. PMID 458883
- [Background] Wu Y, Yin Q, Rui Y, Sun Z, Gu S. Ilizarov technique: Bone transport versus bone shortening-lengthening for tibial bone and soft-tissue defects. J Orthop Sci. 2018 Mar;23(2):341-345. doi: 10.1016/j.jos.2017.12.002. Epub 2017 Dec 28. PMID 29290472
- [Background] Hertel R, Gerber A, Schlegel U, Cordey J, Ruegsegger P, Rahn BA. Cancellous bone graft for skeletal reconstruction. Muscular versus periosteal bed--preliminary report. Injury. 1994;25 Suppl 1:A59-70. doi: 10.1016/0020-1383(94)90263-1. PMID 7927661
- [Background] Tong K, Zhong Z, Peng Y, Lin C, Cao S, Yang Y, Wang G. Masquelet technique versus Ilizarov bone transport for reconstruction of lower extremity bone defects following posttraumatic osteomyelitis. Injury. 2017 Jul;48(7):1616-1622. doi: 10.1016/j.injury.2017.03.042. Epub 2017 Apr 4. PMID 28408083
- [Background] Catagni MA, Azzam W, Guerreschi F, Lovisetti L, Poli P, Khan MS, Di Giacomo LM. Trifocal versus bifocal bone transport in treatment of long segmental tibial bone defects. Bone Joint J. 2019 Feb;101-B(2):162-169. doi: 10.1302/0301-620X.101B2.BJJ-2018-0340.R2. PMID 30700126
- [Background] Zhang Y, Wang Y, Di J, Peng A. Double-level bone transport for large post-traumatic tibial bone defects: a single centre experience of sixteen cases. Int Orthop. 2018 May;42(5):1157-1164. doi: 10.1007/s00264-017-3684-y. Epub 2017 Nov 11. PMID 29129017